CLINICAL TRIAL: NCT02041494
Title: Study Comparing the Efficacy, Safety, and Cost of a Permanent, Synthetic Prosthetic Versus a Biologic Prosthetic in the One-stage Repair of Ventral Hernias in Clean and Contaminated Wounds.
Brief Title: Complex Ventral Hernia Repair Using Biologic or Synthetic Mesh
Acronym: CVHR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Rising costs have made continuing the study untenable
Sponsor: Hobart Harris (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Hobart Harris, Professor, Chief of General Surgery, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCSF-NIDDK-1R21DK093006-01A1; 1R21DK093006-01A1 (NIH)
Record Dates: First submitted 2014-01-18; First posted 2014-01-22 (Estimated); Results first posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-02

CONDITIONS: Hernia, Ventral
Keywords: Hernia; Ventral; Incisional; Abdominal; Herniorrhaphy; Recurrence; Infection; Mesh; Biologic; Synthetic
MeSH Terms: conditions — Hernia, Ventral; Hernia; Surgical Wound; Recurrence; Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Synthetic (Active Comparator): Patients in this arm will have their ventral hernia repaired utilizing Ventralight, a synthetic prosthetic mesh made of polypropylene.
  Interventions: Device: Ventralight
- Biologic (Active Comparator): Patients in this arm will have their ventral hernia repaired utilizing Strattice, a biologic prosthetic mesh derived from porcine dermis.
  Interventions: Device: Strattice

INTERVENTIONS:
Device: Ventralight
  Other Names: Ventralight ST Mesh; K101851
  Arms: Synthetic
Device: Strattice
  Other Names: LTM Surgical Mesh; K070560
  Arms: Biologic

SUMMARY:
Hernias are often treated using a prosthetic mesh to add support to the healing wound. Prosthetic meshes have been used for decades to repair ventral hernias, level 1 data regarding which type of mesh to use is limited. The purpose of this study is to compare the effects, good and/or bad, of two types of prosthetic meshes: one that is made from pig skin (called a "biologic prosthetic"), and one that is made in a laboratory (called a "synthetic prosthetic"). This study will include some patients who have an infection in/near the hernia, and other patients who do not have an infection. We expect the synthetic mesh to be associated with a higher rate of early post-operative surgical site infection and fluid collections (seromas), while we expect the biologic mesh to be associated with a higher rate of recurrence.

DETAILED DESCRIPTION:
This is a prospective, single-blind, randomized study comparing the clinical efficacy and overall costs of two prosthetic meshes in the repair of complex ventral hernias. The two prosthetic meshes to be studied are Ventralight (Bard, Murray Hill, NJ), a synthetic mesh chiefly made of polypropylene and Strattice (LifeCell, Branchburg, NJ), a biologic mesh derived from porcine dermis. The study population will consist of patients who are in need of a repair of a complex ventral hernia. Patients will be enrolled in the study for 24 months following their operation or until they experience a recurrence of their hernia, whichever occurs first. The primary outcome variable is recurrence and the secondary outcome variables are post-operative surgical site infections and overall costs.

There is no universally agreed upon definition of what constitutes a "complex" ventral hernia. For our purposes, a "complex" ventral hernia is one that involves a compromised surgical field, in which gastrointestinal, biliary, or genitourinary procedures are performed, one in which the wound class is considered clean-contaminated, contaminated, or dirty due to other causes, such as infected meshes and enterocutaneous fistulas, or surgical procedures conducted in patients with large ventral hernia defects (>10 cm in any single dimension).

ELIGIBILITY:
Inclusion Criteria:

* Clinical evidence of a midline, ventral hernia, regardless of degree of wound contamination, with the exception of class IV wounds due to the presence/discovery of fecal peritonitis. Specifically, the repair will or will not involve a compromised surgical field in which gastrointestinal, biliary and/or genitourinary procedures will be performed. The surgical wound class may be classified as clean, or it may be classified as clean-contaminated, contaminated, or dirty-infected, due to the repair of an enterocutaneous fistula, takedown of an intestinal stoma and/or removal of infected mesh
* Age >21
* Negative pregnancy test
* No allergic, religious or ethical objections to either polypropylene or porcine prosthetics
* Signed, witnessed informed consent to take part in the study

Exclusion Criteria:

* Lactating women
* Patients who are unable to commit to the follow evaluations over 24 months
* Severe malnutrition (serum albumin <2.0 in the setting of a normal CRP)
* Use of an investigational agent within 1 month prior to study enrollment and/or planned during this study
* Presence of pre-existing parenchymal liver disease characterized by the presence of Child's Class C liver dysfunction (including all of the following: bilirubin ≥ 3.0 mg/dL; albumin ≤ 3.0 mg/dL; refractory ascites; encephalopathy or coma; and poor nutritional status)
* Immunocompromised patients, as evidenced by: administration of high doses of corticosteroids (i.e. doses ≥ 1.5 mg/kg/day of prednisone or equivalent) within 72 hours before study enrollment; status post solid organ transplant or bone marrow transplant and experiencing acute organ rejection or bone marrow failure or rejection; evidence of neutropenia (absolute neutrophil count ≤ 500 cells/mm3 (≤ 500 x 106 cells/L); chemotherapy or radiation therapy within 90 days before study enrollment; known AIDS; any disease sufficiently advanced to suppress resistance to infection (including, but not limited to leukemia, lymphoma or hypogammaglobulinemia); administration of immunoglobulin of G-CSF within 90 days before study enrollment
* Ascites refractory to medical management
* Presence of an underlying disease/injury with life expectancy less than two years and/or severe underlying disease that would preclude study entry (e.g. known malignancy)
* Wound Classification IV due to the presence/discovery of fecal peritonitis. Other cases of wound class IV including presence of purulent inflammation, soft tissue/mesh infection, or visceral perforation resulting in a contained fistula (e.g. enterocutaneous fistula) are still considered eligible for enrollment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hobart W. Harris, M.D., M.P.H., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Harris HW, Primus F, Young C, Carter JT, Lin M, Mukhtar RA, Yeh B, Allen IE, Freise C, Kim E, Sbitany H, Young DM, Hansen S. Preventing Recurrence in Clean and Contaminated Hernias Using Biologic Versus Synthetic Mesh in Ventral Hernia Repair: The PRICE Randomized Clinical Trial. Ann Surg. 2021 Apr 1;273(4):648-655. doi: 10.1097/SLA.0000000000004336. PMID 33443907

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adults (≥21 years of age) with a ventral hernia scheduled for an elective repair were eligible for inclusion. Recruitment and all surgical procedures were carried out from March 2014 through October 2018 at UCSF Medical Center). All participants were recruited via referral to the medical center's surgery clinics. Patients were only enrolled once.
Groups:
- Biologic: Patients in this arm will have their ventral hernia repaired utilizing Strattice, a biologic prosthetic mesh derived from porcine dermis.
  Strattice
- Synthetic: Patients in this arm will have their ventral hernia repaired utilizing a synthetic prosthetic mesh made of polypropylene.
  SoftMesh/Ventralight ST
Period: Overall Study
Arm/Group | Biologic | Synthetic
Started | 82 | 83
Completed | 63 | 63
Not Completed | 19 | 20
Not completed — Death | 1 | 3
Not completed — Lost to Follow-up | 2 | 6
Not completed — study terminated | 16 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synthetic | Biologic | Total
Number analyzed (Participants) | 83 | 82 | 165
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.5 (11.1) | 55.0 (11.5) | 55.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 47 | 97
  Male | 33 | 35 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 4 | 5 | 9
  White | 59 | 50 | 109
  More than one race | 4 | 3 | 7
  Unknown or Not Reported | 14 | 21 | 35
Region of Enrollment [Number; unit: participants]
  United States | 83 | 82 | 165

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Had a Recurrence of Hernia, at Anytime, up to Two Years Following Repair.
Description: Number of patients who had a recurrence of hernia, at anytime, up to two years following repair as determined by physical examination, ultrasound or CT scan.
Time Frame: up to 24 months after surgery
Population: This measure includes patients that recurred before 2 years and were not followed for 2 years, and some patients that recurred were followed for 2 years.
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic | Synthetic
Number analyzed (Participants) | 63 | 64
Participants | 25 | 14

2. Secondary Outcome: Number of Patients Who Experienced Surgical Site Infections.
Description: Number of patients who experienced surgical site infections as determined by physical examination.
Time Frame: 30 days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Biologic | Synthetic
Number analyzed (Participants) | 82 | 83
Participants | 32 | 28

3. Other Pre Specified Outcome: Generic Measure of Health-related Quality of Life and Hernia-specific Measure of Quality of Life With a Focus on Abdominal Wall Function
Description: Quality of life will be measured using the SF-36 and the HerQLes surveys.
Time Frame: 24 months after surgery
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Number of Surgical Site Occurrences
Description: Number of surgical site occurrences by type.
Time Frame: Up to two years from surgery
Population: Only patients with a surgical site occurrence were included in this outcome measure.
Measure: Number; unit: surgical site occurence
Groups:
- Synthetic: Patients in this arm will have their ventral hernia repaired utilizing Ventralight, a synthetic prosthetic mesh made of polypropylene.
  Ventralight
Arm/Group | Biologic | Synthetic
Number analyzed (Participants) | 17 | 18
surgical site occurence
  Hematoma: number analyzed (Participants) | 4 | 0
  Hematoma | 5 |
  Seroma: number analyzed (Participants) | 6 | 10
  Seroma | 7 | 12
  Wound necrosis and other: number analyzed (Participants) | 7 | 8
  Wound necrosis and other | 9 | 10

5. Other Pre Specified Outcome: Number of Other Surgical Complications
Description: Number of other surgical complications including: urinary tract infections, pneumonia, and Deep Vein Thrombosis/pulmonary embolism.
Time Frame: 30 days after surgery
Population: Only patients with other surgical complications were included in this outcome measure.
Measure: Number; unit: occurence
Arm/Group | Biologic | Synthetic
Number analyzed (Participants) | 20 | 13
occurence
  Urinary tract infection: number analyzed (Participants) | 11 | 8
  Urinary tract infection | 13 | 7
  Pneumonia: number analyzed (Participants) | 3 | 1
  Pneumonia | 4 | 1
  Deep Vein Thrombosis/pulmonary embolism: number analyzed (Participants) | 6 | 6
  Deep Vein Thrombosis/pulmonary embolism | 7 | 5

6. Other Pre Specified Outcome: Activity Level
Description: Activity level will be measured using the Activity Assessment Scale.
Time Frame: 24 months after surgery
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Overall Cost
Description: Overall costs will be measured using a combination approach comparing actual costs, allowed vs. paid amounts, and Medicare payment rates using diagnosis related groups (DRG) and resource-based relative value scale (RBRVS) data.
Time Frame: 24 months after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected throughout the duration of the study, an average of 26 months.
Arm/Group | Biologic | Synthetic
All-Cause Mortality (participants affected / at risk) | 0/82 | 2/83
Serious Adverse Events (participants affected / at risk) | 15/82 | 20/83
Other Adverse Events (participants affected / at risk) | 27/82 | 19/83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biologic (N=82) | Synthetic (N=83)
deep space infection (Infections and infestations) | 15 (15) | 19 (19)
death (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Biologic (N=82) | Synthetic (N=83)
superficial SSI (Infections and infestations) | 17 (17) | 9 (9)
urinary tract infection (Renal and urinary disorders) | 11 (11) | 7 (7)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
DVT/pumonary embolism (Blood and lymphatic system disorders) | 6 (6) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2014-07-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT02041494/SAP_000.pdf
  • Study Protocol (2014-07-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT02041494/Prot_001.pdf